CLINICAL TRIAL: NCT00827814
Title: Effect of Dutasteride on Bladder Wall Hypertrophy in Patients With Benign Prostatic Obstruction: A 24-Week Open-Label, Single-Arm Pilot Study
Brief Title: Effect of Dutasteride on Bladder Wall Hypertrophy in Patients With Benign Prostatic Obstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Kyu-Sung Lee/Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-06-022
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Last update posted 2009-06-11 (Estimated); Status verified 2009-06

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dutasteride (Experimental)
  Interventions: Drug: Dutasteride

INTERVENTIONS:
Drug: Dutasteride — Dutasteride 0.5 mg od.
  Other Names: Avodart

SUMMARY:
Increased bladder mass occurs as a consequence of bladder outlet obstruction in animals and patients, and relief of bladder outlet obstruction reverses an increased bladder mass. Whether increased bladder mass is not only a consequence of bladder outlet obstruction but also a relevant risk factor for the progression of lower urinary tract symptoms associated with benign prostate hyperplasia cannot be decided due to a lack of appropriate data, most likely because bladder wall thickness is not routinely measured in clinical studies and/or routine clinical practice. Despite this lack of data, many urologists feel that increased bladder mass should be prevented or decreased to reduce the occurrence of serious complications.

The possibility of using bladder wall thickness data as criteria for benign prostate hyperplasia intervention and as outcome criteria for benign prostate hyperplasia treatment has been proposed. Detrusor hypertrophy associated with bladder outlet obstruction can be imaged on suprapubic ultrasound, and bladder mass can be quantified from the evaluation of bladder wall thickness and bladder volume. Bladder wall hypertrophy has been found to be correlated with detrusor function.

Independent studies have shown that surgical treatment of benign prostatic obstruction results in a significant decrease of bladder mass. Preliminary data suggest the possibility that medical treatment with alpha-adrenergic antagonists might also produce a reduction of bladder wall hypertrophy.

The investigators assume that the prevention of benign prostate hyperplasia progression by alpha-adrenergic antagonists and 5 alpha reductase inhibitors may be result of bladder function protection. To our knowledge there have been no studies that evaluated the effects of a 5 alpha reductase inhibitors on bladder function. Therefore, the investigators plan to conduct a prospective trial evaluating the effects of 5 alpha reductase inhibitors on bladder function by the evaluation of bladder wall thickness and lower urinary tract symptoms.

DETAILED DESCRIPTION:
1 Objective

1.1 Primary Objective: To explore the efficacy of Dutasteride in reducing bladder wall hypertrophy from baseline to 6 months of treatment in male patients with benign prostatic obstruction.

1.2 Secondary Objective:

1. To explore the efficacy of Dutasteride in reducing the LUTS symptoms, number of micturitions, and number of urgency episodes from baseline to 6 months of treatment
2. To explore the efficacy of Dutasteride on the urodynamic parameters from baseline to 6 months of treatment.
3. To explore the efficacy of Dutasteride on the tolerability, safety, patient perception and quality of life from baseline to 6 months of treatment.

2 Endpoints

2.1 Primary Endpoint: Percent (numeric) changes in ultrasound-estimated bladder weight (UEBW) from baseline to 6 months of treatment

2.2 Secondary Endpoint:

Urodynamic parameters: From baseline to 6 months of treatment

• Percentage and numeric changes of the

* Maximum flow rate (mL/s)
* Average flow rate (mL/s)
* Post-void residual urine volume (mL)

Micturition diary efficacy parameters: From baseline to 6 months of treatment

* Percentage and numeric changes in micturition frequency/24 hours
* Percentage and numeric changes in mean volume voided per micturition
* Percentage and numeric changes in mean number and severity of urgency per micturition

Prostate volume parameters:

• Change in prostate volume by TRUS from baseline to after 6 months of treatment.

• Change in serum PSA from baseline to after 6 months of treatment.

Quality of life parameters:

• Change in Bother Score of IPSS score from baseline to 6 months of treatment

LUTS Symptom parameters:

• Change in IPSS score from baseline to 6 months of treatment

- total score: sum of all 7 questions

* storage score: sum of questions 2, 4 and 7
* voiding score: sum of questions 1, 3, 5 and 6

LUTS outcome score (LOS)

• Change in LOS from baseline to 6 months of treatment

Patient perceptions:

* Patient perception of treatment benefit after 3 and 6 months of treatment
* Change in patient perception of urgency from baseline to 3 and 6 month of treatment

Safety parameters:

• Incidence and severity of adverse events

• Incidence and reason of withdrawals

3. STUDY DESIGN AND METHODS

Study Design: This is a 6-month prospective Phase IV study to explore the effect on the bladder function of Dutasteride in male patients with benign prostatic obstruction.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥50 and <80 years old
2. Presence of LUTS for at least 3 months
3. IPSS≥15
4. Bladder outlet obstruction confirmed by pressure-flow study (BOOI > 20)
5. Prostate volume measured by TRUS ≥ 30ml and < 100ml
6. Able to comply with the prescribed treatment protocol and evaluations.

Exclusion Criteria:

1. Patients with neurogenic voiding disorders
2. Patients with prostate or bladder cancer
3. Patients underwent urethral, prostate or bladder neck surgery
4. Patients with urethral stricture or bladder neck contracture
5. Serum PSA≥4ng/ml (if the patient confirmed as no malignancy by prostate biopsy can be included).
6. Patients who medicated with 5ARI within 6 months
7. Patients who do not agree with the informed consent

Ages: 50 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-06; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Percent (numeric) changes in ultrasound-estimated bladder weight (UEBW) | Baseline and 6 months of dutasteride treatment

SECONDARY OUTCOMES:
Urodynamic parameters | Baseline and 3 and/or 6 months of dutasteride treatment
Micturition diary efficacy parameters | Baseline and 3 and/or 6 months of dutasteride treatment
Prostate volume parameters | Baseline and 3 and/or 6 months of dutasteride treatment
Quality of life parameters | Baseline and 3 and/or 6 months of dutasteride treatment
LUTS Symptom parameters | Baseline and 3 and/or 6 months of dutasteride treatment
LUTS outcome score | Baseline and 3 and/or 6 months of dutasteride treatment
Patient perceptions | Baseline and 3 and/or 6 months of dutasteride treatment
Safety parameters | Baseline and 3 and/or 6 months of dutasteride treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Lee, Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea